CLINICAL TRIAL: NCT04500028
Title: Clinical Outcomes of Vaginal Isonicotinic Acid Hydrazide (INH) Administration Prior to Levonorgestrel Releasing Intrauterine System Insertion in Women Delivered Only by Elective Cesarean Section: a Randomized Double Blinded Clinical Trial
Brief Title: Vaginal Isonicotinic Acid Hydrazide Administration Prior to Insertion Levonorgestrel-releasing Intrauterine System
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, A Professor, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/355/3/19
Record Dates: First submitted 2020-08-02; First posted 2020-08-05 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: IUCD Complication

STUDY DESIGN:
Intervention Model Description: double blind randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INH (Experimental): 3 vaginal tablet of isonicotinic acid hydrazide (900mg) ( inserted by the study nurse 4 hours before IUD insertion.
  Interventions: Drug: INH
- Placebo Comparator (Placebo Comparator): one tablet of placebo inserted by the study nurse 4 hours before IUD insertion.
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: INH — 3 vaginal tablet of isonicotinic acid hydrazide (900mg) inserted by the study nurse 4 hours before IUD insertion.
  Arms: INH
Drug: Placebo Comparator — 3 tablet of placebo inserted by the study nurse 4 hours before IUD insertion.
  Arms: Placebo Comparator

SUMMARY:
To investigate whether vaginal isonicotinic acid hydrazide (INH) administered before the levonorgestrel-releasing intrauterine system(IUs) insertion reduces failed insertions, insertion-related complications, and pain in Women With no Previous Vaginal Delivery.

DETAILED DESCRIPTION:
Long-acting reversible contraception methods are highly effective methods for reduction of the unplanned pregnancy rate worldwide. The intrauterine device is a single procedure that provides reliable, effective and long term contraception for many women. However, the insertion procedure can be associated with a troublesome degree of pain that prevent some women from choosing its use. Different interventions have been described to decrease pain perception during intrauterine device insertion with no agreement on an effective one.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant women
* Women that did not receive any analgesics or Dinoprostone in the 24 hours prior to insertion
* Women who delivered only by cesarean section

Exclusion Criteria:

* Women with any uterine abnormalities such as congenital anomalies, endometrial lesions, adenomyosis, or fibroids.
* Those with a Category 3 or 4 conditions for intrauterine device insertion according to the WHO Medical Eligibility Criteria for contraceptive use
* Allergy to isonicotinic acid hydrazide
* known psychiatric disorders ( anxiety and depression) and chronic use of medications that could interfere with pain perception (antidepressants and anticonvulsants)
* Women refuse to participate in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Non-pregnant women who delivered only by cesarean section
Enrollment: 220 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
The difference in pain scores during intrauterine device insertion | 10 minutes
  The difference in pain scores during intrauterine device insertion using visual analog scale from 0 to 10

SECONDARY OUTCOMES:
duration of IUD insertion | 10 minutes
  duration of IUD insertion measured in minutes

CONTACTS AND LOCATIONS:
Overall Officials: nahla w Shady, md, Study Chair — Aswan universirty
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No